CLINICAL TRIAL: NCT00005648
Title: A Phase III, Double-Blind, Placebo Controlled Trial of Gemcitabine Plus Placebo Versus Gemcitabine Plus R115777 in Patients With Advanced Pancreatic Cancer
Brief Title: Gemcitabine With or Without Tipifarnib (R115777) in Treating Patients With Advanced Pancreatic Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sr Dir Clinical Research, Johnson & Johnson Pharmaceutical Research and Development, L.L.C.
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CR003976; R115777-INT-11
Record Dates: First submitted 2000-05-02; First posted 2004-05-21 (Estimated); Last update posted 2011-05-19 (Estimated); Status verified 2010-10

CONDITIONS: Pancreatic Neoplasms
Keywords: Stage II pancreatic cancer; Stage III pancreatic cancer; Recurrent pancreatic cancer; Adenocarcinoma of the pancreas; Stage IV pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine; tipifarnib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- 001 (Experimental): Gemcitabine with R115777 R115777 200 mg oral twice daily at 12-hour intervals throughout the study coadministered with gemcitabine 1000 mg/m2 iv every week for the first 7 weeks followed by 1 week rest and then every 3 out of 4 weeks thereafter for up to 5 years
  Interventions: Drug: Gemcitabine with R115777
- 002 (Placebo Comparator): Gemcitabine with Placebo Placebo oral twice daily at 12-hour intervals throughout the study coadministered with gemcitabine 1000 mg/m2 iv every week for the first 7 weeks followed by 1 week rest and then every 3 out of 4 weeks thereafter for up to 5 years
  Interventions: Drug: Gemcitabine with Placebo

INTERVENTIONS:
Drug: Gemcitabine with R115777 — R115777 200 mg, oral, twice daily at 12-hour intervals throughout the study coadministered with gemcitabine, 1000 mg/m2, iv, every week for the first 7 weeks, followed by 1 week rest, and then every 3 out of 4 weeks thereafter for up to 5 years
  Arms: 001
Drug: Gemcitabine with Placebo — Placebo, oral, twice daily at 12-hour intervals throughout the study coadministered with gemcitabine, 1000 mg/m2, iv, every week for the first 7 weeks, followed by 1 week rest, and then every 3 out of 4 weeks thereafter for up to 5 years
  Arms: 002

SUMMARY:
The purpose of this study is to compare the effectiveness of gemcitabine with or without tipifarnib (R115777) in patients who have advanced pancreatic cancer.

DETAILED DESCRIPTION:
This is a randomized (study drug assigned by chance), double-blind (neither the investigator or patient will know the identity of the assigned treatment) to compare the overall survival of patients with advanced pancreatic cancer after treatment with gemcitabine with and without tipifarnib (referred to as R115777). Gemcitabine is an approved chemotherapy agent administered intravenously (iv) (though a vein) for patients with advanced pancreatic cancer. R115777 is an orally (by mouth) administered investigational drug that is being tested in combination with gemcitabine for the treatment of patients with advanced pancreatic cancer. Patients will continue to receive treatment with gemcitabine and R115777 (or placebo) unless disease progression or unacceptable toxicity is observed. All patients in the study will be followed for study assessments and safety for up to the 5 years, the start of further treatment, or death (whichever comes first). R115777 (or matching placebo) 200 mg will be orally administered at intervals of approximately 12 hours daily throughout the study. Gemcitabine will be administered iv at a starting dose of 1000 mg/m2 every week for the first 7 weeks, followed by 1 week rest, and then every 3 out of 4 weeks thereafter. Treatment with gemcitabine and tipifarnib (or placebo) will continue for up to 5 years (or until the start of further treatment) in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Pathological (confirmed by biopsy) diagnosis of pancreatic cancer
* have an Eastern Cooperative Oncology Group (ECOG) performance score of 0 to 1 (defined as a patient who does not have symptoms of pancreatic cancer and is fully active or who has symptoms but is able to light work)

Exclusion Criteria:

* Have absolute neutrophil (white blood cell) count, platelet count (blood clotting factors), or results from liver function tests considered by the investigator to be significantly abnormal
* Newly diagnosed disease that has the potential for curative surgical resection
* Prior therapy with any chemotherapy, or any other systemic therapy for pancreatic cancer
* Have cardiovascular disease considered by the investigator to be uncontrolled or severe

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 688 (Actual)
Dates: Start 1999-11; Study Completion 2003-11 (Actual)

PRIMARY OUTCOMES:
Overall survival of patients with advanced pancreatic cancer after treatment with gemcitabine with or without R115777. | From the date of randomization to the date of death or to the last followup date for patients who were still alive at the clinical cutoff date (ie, for up to 5 years)

SECONDARY OUTCOMES:
Evaluation of Quality of Life (QOL) parameters in patients with advanced pancreatic cancer after treatment with gemcitabine with or without R115777 | From the date of randomization to the date of death or to the last followup date for patients who were still alive at the clinical cutoff date (ie, for up to 5 years)
The incidence of adverse events with respect to severity and relationship to the study medication as a measure of safety | From the date of randomization to the date of death or to the last followup date for patients who were still alive at the clinical cutoff date (ie, for up to 5 years)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- See also: Gemcitabine With or Without tipifarnib (R115777) in Treating Patients With Advanced Pancreatic Cancer — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=548&filename=CR003976_CSR.pdf